CLINICAL TRIAL: NCT04085809
Title: A 14-Day, Single-Blind, Controlled Study to Assess the Qualitative Improvement in Skin Moisturization and Desquamation of AmLactin® Rapid Relief Treatment in Healthy Female Subjects
Brief Title: This Was a Clinical Study Investigating the Moisturization and Desquamation Effect of AmLactin® Rapid Relief Restoring Lotion + Ceramides on Dry Skin in Healthy Female Volunteers. AmLactin® Rapid Relief is an Over-the-counter Cosmetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0123-02-01
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Dry Skin

STUDY DESIGN:
Intervention Model Description: Upon enrollment, each subject received a randomization code, indicating which leg the study product had to be applied (the other leg received no study product). Each subject in this study served as her own control.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Leg: AmLactin® Rapid Relief / Right Leg: No Treatment (Experimental): AmLactin® Rapid Relief, BID application for 14 days on left leg and no treatment on right leg
  Interventions: Other: AmLactin® Rapid Relief
- Left Leg: No Treatment / Right Leg: AmLactin® Rapid Relief (Experimental): AmLactin® Rapid Relief, BID application for 14 days on right leg and no treatment on left leg
  Interventions: Other: AmLactin® Rapid Relief

INTERVENTIONS:
Other: AmLactin® Rapid Relief — AmLactin® Rapid Relief, BID application for 14 days. AmLactin is an over-the-counter cosmetic.

SUMMARY:
The primary objective of this study was to investigate if AmLactin® Rapid Relief improves the skin through desquamation and moisturization via D-SQUAME analysis. AmLactin® Rapid Relief is an over-the-counter cosmetic.

ELIGIBILITY:
Inclusion Criteria:

* healthy female (confirmed by medical history) with Fitzpatrick skin types I-VI
* dry, rough skin on the anterior shins (defined as Grade 3-4 on the dermatologist evaluation of the skin);

Exclusion Criteria:

- Had any visible skin disease at the assessment site which, in the opinion of the Investigator, would interfere with the evaluation of the test site

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants were being studied
Enrollment: 56 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in D-SQUAME | Baseline, Day 2, Day 14
  D-SQUAME is a sticky tape that is placed on the skin and the more skin that comes off on the tape, the drier the skin and less moisturization and desquamation.

SECONDARY OUTCOMES:
Change from baseline in overall dry skin scale | Baseline, Day 2, Day 14
  An evaluation of the skin by a blinded Investigator was utilized to assess the overall appearance of the skin on an ordinal scale from 0 = none to 4 = severe in five domains.
Change from baseline in Skin Dryness assessed by Dry Skin Scale | Baseline, Day 2, Day 14
  An evaluation of the skin by a blinded Investigator was utilized to assess the overall appearance of the skin on an ordinal scale from 0 = none to 4 = severe.
Change from baseline in Skin Texture/Roughness (Tactile) assessed by Dry Skin Scale assessed by Dry Skin Scale | Baseline, Day 2, Day 14
  An evaluation of the skin by a blinded Investigator was utilized to assess the overall appearance of the skin on an ordinal scale from 0 = none to 4 = severe.
Change from baseline in Skin Texture/Roughness (Visual) assessed by Dry Skin Scale | Baseline, Day 2, Day 14
  An evaluation of the skin by a blinded Investigator was utilized to assess the overall appearance of the skin on an ordinal scale from 0 = none to 4 = severe.
Change from baseline in Desquamation/Flakiness assessed by Dry Skin Scale | Baseline, Day 2, Day 14
  An evaluation of the skin by a blinded Investigator was utilized to assess the overall appearance of the skin on an ordinal scale from 0 = none to 4 = severe.
Change from baseline in Luminosity/Radiance assessed by Dry Skin Scale | Baseline, Day 2, Day 14
  An evaluation of the skin by a blinded Investigator was utilized to assess the overall appearance of the skin on an ordinal scale from 0 = none to 4 = severe.
Change from baseline in Subject Self-Assessment Questionnaire | Baseline, Day 14
  Subjects rated the skin attributes of the treated leg in nine domains on a scale from 0 - 4 .

CONTACTS AND LOCATIONS:
Locations (1):
- Sandoz Investigational Site, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Draelos ZD, Hall S, Munsick C. A 14-day Controlled Study Assessing Qualitative Improvement with 15% Lactic Acid and Ceramides in Skin Moisturization and Desquamation. J Clin Aesthet Dermatol. 2020 Aug;13(8):E54-E58. Epub 2020 Aug 1. PMID 33178384